CLINICAL TRIAL: NCT05243875
Title: Lupus Education Alliance Program
Acronym: LEAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early Termination
Sponsor: Tulane University (Other)
Collaborators: University of Alabama at Birmingham (Other); Ochsner Health System (Other); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, David Chae, Associate Professor, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00073870
Record Dates: First submitted 2021-11-15; First posted 2022-02-17 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus; COVID-19
MeSH Terms: conditions — Lupus Erythematosus, Systemic; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a two-arm study in which participants are randomized to an experimental (education + navigation) or comparison (education only) group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education / Navigation (Experimental): COVID education involving providing information about COVID for people with SLE and CDC recommendations for testing, testing options (e.g., pharmacies, doctors' offices, at-home), treatment in the event of a positive COVID result, and current recommendations around vaccination for those with SLE; and (2) navigation, which involves individual tailoring of information about where and how to get tested, and where to get vaccinated, and when appropriate, guiding participants in scheduling testing and vaccination appointments.
  Interventions: Behavioral: LEAP Education + Navigation
- Education Only (Active Comparator): COVID education involving providing information about COVID for people with SLE and CDC recommendations for testing, testing options (e.g., pharmacies, doctors' offices, at-home), treatment in the event of a positive COVID result, and current recommendations around vaccination for those with SLE.
  Interventions: Behavioral: LEAP Education

INTERVENTIONS:
Behavioral: LEAP Education + Navigation — COVID education involving providing information about COVID for people with SLE and CDC recommendations for testing, testing options (e.g., pharmacies, doctors' offices, at-home), treatment in the event of a positive COVID result, and current recommendations around vaccination for those with SLE; and (2) navigation, which involves individual tailoring of information about where and how to get tested, and where to get vaccinated, and when appropriate, guiding participants in scheduling testing and vaccination appointments.
  Arms: Education / Navigation
Behavioral: LEAP Education — COVID education involving providing information about COVID for people with SLE and CDC recommendations for testing, testing options (e.g., pharmacies, doctors' offices, at-home), treatment in the event of a positive COVID result, and current recommendations around vaccination for those with SLE.
  Arms: Education Only

SUMMARY:
Randomized controlled trial of a COVID-19 behavioral and educational intervention for people with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
Randomized controlled trial of a COVID-19 behavioral and educational intervention for people with systemic lupus erythematosus (SLE).

ELIGIBILITY:
18 years or older, ability to understand and speak English, diagnosis of SLE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of COVID testing | 3 months
  Participant-reported COVID testing
Incidence of COVID-19 Vaccination | 3 months
  Participant-reported COVID vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to researchers outside the study team after completion of the primary analyses. Data requests, including a list of variables and analytic plan, will be sent to the Project Coordinator and reviewed by the PI, who will approve or deny the data request.